CLINICAL TRIAL: NCT02310776
Title: Breast Lesion Detection Using the Acuson S2000 Automated Breast Volume Scanner (ABVS) Compared With Handheld (HH) Physician-performed Ultrasound (US) Examinations
Brief Title: Lesion Detection of Automated Breast Ultrasound Compared With Handheld Physician-performed Breast Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Ellen Mendelson, MD, FACR, Lee F. Rogers Professor of Medical Education in Radiology, Professor of Radiology Feinberg School of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00043696
Record Dates: First submitted 2014-11-25; First posted 2014-12-08 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Automated & Handheld breast US exams (Other): 1. Automated breast ultrasound exam: 3D supine automated breast ultrasound scanner.
  2. Handheld breast ultrasound exam: High-resolution handheld breast ultrasound.
  Interventions: Device: Supine automated breast ultrasound scanner; Device: High-resolution handheld breast ultrasound

INTERVENTIONS:
Device: Supine automated breast ultrasound scanner — Automated wide-field-of-view breast ultrasound volume scan performed by a sonographer and interpreted by a breast imaging radiologist.
Device: High-resolution handheld breast ultrasound — Standard of care, small field-of-view 2D breast ultrasound performed and interpreted by a breast imaging radiologist

SUMMARY:
Compare lesion detection of the automated breast ultrasound (ABVS) exam with the conventional handheld (HH) breast ultrasound (US) exam.

DETAILED DESCRIPTION:
This is a research study to test a FDA-approved automated breast ultrasound (ABVS) machine in subjects recommended for an ultrasound of the breast. The main purpose of the study is to compare images obtained from the automated breast ultrasound exam with the standard physician performed handheld breast ultrasound exam for lesion detection equivalence.

Each subject will have a bilateral hand-held breast ultrasound and a bilateral automated breast ultrasound, both exams preferably done on the same day. The hand-held ultrasound will be performed by a breast imaging physician participating in the study and the automated ultrasound exam will be performed by a sonographer.

There is no radiation risk from ultrasound. The physician performing the handheld breast ultrasound is blinded to the study, will not know the subject's history, but only the reason for the breast ultrasound exam.

The automated scan requires gentle pressure on the breast during a scan. Three basic views will be acquired for each breast, each scan lasting approximately one minute. Once all necessary views are acquired, the images will be sent to a remote workstation, where a second radiologist, also blinded to the results of the handheld study, will interpret the automated ultrasound.

Once all images and patient information are gathered, the study radiologists will review the previous images, if available, to provide the final result that will determine clinical management. Therefore, it is possible that the hand-held or automated ultrasound scan will lead to further evaluation of the breast and possibly a biopsy.

ELIGIBILITY:
Inclusion Criteria:

* anyone who is referred for an ultrasound of the breast

Exclusion Criteria:

* Subjects whose breast thickness is greater than 6 cm.The maximum depth of image filed for the ABVS acquisition is 6 cm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen B Mendelson, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Medicine, Chicago, Illinois
  - Weinstein Imaging, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Automated & Handheld Breast US Exams: 1. Automated breast ultrasound exam: 3D supine automated breast ultrasound scanner; Supine automated breast ultrasound scanner: Automated wide-field-of-view breast ultrasound volume scan performed by a sonographer and interpreted by a breast imaging radiologist.
  2. Handheld breast ultrasound exam: High-resolution handheld breast ultrasound; Standard of care, small field-of-view 2D breast ultrasound performed and interpreted by a breast imaging radiologist
Period: Overall Study
Arm/Group | Automated & Handheld Breast US Exams
Started | 501
Completed | 501
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Automated & Handheld Beast US Exams: 1. Automated breast ultrasound exam: 3D supine automated breast ultrasound scanner; Supine automated breast ultrasound scanner: Automated wide-field-of-view breast ultrasound volume scan performed by a sonographer and interpreted by a breast imaging radiologist.
  2. Handheld breast ultrasound exam: High-resolution handheld breast ultrasound; Standard of care, small field-of-view 2D breast ultrasound performed and interpreted by a breast imaging radiologist
Arm/Group | Automated & Handheld Beast US Exams
Number analyzed (Participants) | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 461
  >=65 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 501
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 501

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Lesions Detected With Automated Breast Ultrasound (ABVS) Compared to the Standard of Care Handheld (HH) Breast Ultrasound (US)
Description: Solid lesions found on whole breast 3D supine automated breast ultrasound are compared in number and identity with solid lesions found using high resolution standard of care handheld breast ultrasound performed by physicians
Time Frame: Time for performance of ABVS was measured separately from interpretation time. Time for performance of real time HH whole breast US was also measured. For HH US physician performed, performance included interpretation.
Population: Each participant was evaluated based on Breast Imaging-Reporting and Data System (BI-RADS) assessment for Automated and Handheld breast ultrasound exams. If participant had more than one lesion, each lesion was assessed and listed separately and if a participant did not have a lesion, she was entered once.
Measure: Number (95% Confidence Interval); unit: Detection ratio of lesions
Units Other Than Participants: Lesions
Arm/Group | Automated & Handheld Breast US Exams
Number analyzed (Participants) | 501
Number analyzed (Lesions) | 744
Detection ratio of lesions | 1.19 [1.06 to 1.34]

ADVERSE EVENTS:
Arm/Group | Automated & Handheld Breast US Exams
Serious Adverse Events (participants affected / at risk) | 0/501
Other Adverse Events (participants affected / at risk) | 0/501

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No